CLINICAL TRIAL: NCT04221997
Title: Extracellular Vesicles as Predictors of Antidepressant Outcomes in Pediatric Anxiety (EV-SOPRANO)
Brief Title: Trial With the Treatment of Sertraline in Youth With Generalized, Separation and/or Social Anxiety Disorders.
Acronym: EV-SoPRANO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jeffrey Strawn, MD, Associate professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Strawn EV-SoPRANO; R01HD098757 (NIH)
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Sertraline

STUDY DESIGN:
Intervention Model Description: During the acute treatment phase, 90 patients will be randomized to sertraline and 30 patients will be randomized to placebo (3:1).
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- sertraline (Experimental): 90 patients will be randomized to sertraline
  Interventions: Drug: sertraline
- Placebo (Placebo Comparator): 30 patient will be randomized to placebo
  Interventions: Drug: sertraline
- Healthy Control (No Intervention): 30 healthy comparison subjects will be followed over the course of 12 weeks

INTERVENTIONS:
Drug: sertraline — Sertraline is an antidepressant in a group of drugs called selective serotonin reuptake inhibitors (SSRIs)
  Other Names: Zoloft
  Arms: Placebo; sertraline

SUMMARY:
A Multicenter, acute, randomized, double-blind, placebo-controlled, flexible-dose trial with the treatment of sertraline.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled trial of an evidence-based antidepressant, sertraline, in youth (N=120) with generalized, separation and/or social anxiety disorders, seeks to evaluate the predictive value of plasma EV signatures. Patients will be randomized to sertraline (25-200 mg/day) or placebo (3:1) and total plasma EVs will be collected at baseline and serially during the course of the 12-week treatment period.

ELIGIBILITY:
Inclusion Criteria for Patients with Anxiety :

* Written, informed assent and consent.
* Patients, parent/guardian/LAR must be fluent in the English.
* 8-17 years of age, inclusive, at Visit 1, and who have a parent/guardian/LAR.
* Patients must meet DSM-5 criteria for generalized, social and/or separation anxiety disorder, confirmed by the MINI-KID with no lifetime history of mania, OCD or significant history of trauma exposure.
* PARS score ≥15 at Visits 1 and 2.
* Caregiver who is willing to consent to be responsible for safety monitoring of the patient, provide information about the patient's condition, oversee the administration of the investigational product.
* No clinically significant abnormalities on physical examination.
* Negative pregnancy test at Visit 1 in females.
* Sexually active patients must practice a reliable method of contraception (Section 15.0) that will continue for the duration of the study and within 30 days following the end of study participation.
* Reliable methods of contraception are defined below; other forms of contraceptives (pharmacological and/or non-pharmacological) are not accepted.

  * surgical sterilization
  * oral contraceptives (e.g., estrogen-progestin combination or progestin)
  * transdermally-delivered contraceptives (e.g., Ortho-Evra), depot injections (e.g.,
  * Depo-Provera)
  * vaginal contraceptive ring (e.g., NuvaRing), contraceptive implants (e.g., Implanon, Norplant
  * II/Jadelle)
  * an intrauterine device or
  * diaphragm plus condom.

Inclusion Criteria for Healthy Controls:

* Written, informed assent and consent.
* Patients, parent/guardian/LAR must be fluent in the English.
* 8 to 17 years of age, inclusive, at Visit 1, and who have a parent/guardian/LAR.
* No history of any DSM-5 disorders (nicotine use disorder is permitted, history of adjustment disorder is permitted), confirmed by the MINI-KID.
* Caregiver who is willing to consent to be responsible for safety monitoring of the patient, provide information about the patient.
* No clinically significant abnormalities on physical examination. Negative pregnancy test at Screening in females.
* Negative urine drug screen at Screening.
* No first-degree relatives with an affective, anxiety or psychotic disorder.

Exclusion Criteria for Patients with Anxiety Disorders and Healthy Comparison:

* Subjects Co-occurring DSM-5 diagnosis mood (except persistent depressive disorder, unspecified depressive disorder or co- occurring anxiety disorders, provided that the primary diagnosis is generalized, social and/or separation anxiety disorder(s)), eating, bipolar, or psychotic disorders.
* A history of treatment with SSRIs within 12 weeks of Visit 2 (Baseline) or current pharmacotherapy with CNS effects that require >5 half-lives for discontinuation.
* A history of major neurological or medical illness or head trauma with loss of consciousness for ≥5 minutes.
* Lifetime history of mania, OCD, or significant history of trauma exposure.
* History of hypersensitivity to sertraline.
* Lifetime diagnosis of intellectual disability or history of IQ <70.
* History of alcohol/substance use disorder or any substance abuse within the past 6 months (nicotine dependence is permitted).
* Current psychotherapy stable for <2 months prior to Visit 2 (Baseline).
* Females will not be eligible to participate if they are pregnant, breast feeding or lactating.
* The subject lives >100 miles from the University of Cincinnati or >90 minutes from the CU site or is not able to attend the follow-up visits.
* Patients who are unable to swallow capsules.
* Is currently considered at risk of suicide in the opinion of the investigator, represents an inappropriate risk to the participant and/or could confound the interpretation of the study results.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Clinical Global Impression-Improvement Scale ≤ 2 | Week 12
  Primary response outcome will be treatment response based on patients having attained a score on the Clinical Global Impression-Improvement Scale ≤ 2 at Week 12 or Last-Observation-Carried-Forward (LOCF).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Strawn, MD, FAACAP, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No